CLINICAL TRIAL: NCT00208702
Title: Thyroid Axis in Major Depression
Brief Title: Thyroid Medication and Antidepressants for Treating Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Boadie W. Dunlop, Director, Mood and Anxiety Disorders Program, Emory University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-1996; R01MH056946 (NIH); 431-1996; DSIR AT-SO
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Major Depression
Keywords: Major Depressive Disorder; Mental Health; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Psychological Well-Being; Depression | interventions — Triiodothyronine; Sertraline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sertraline + triiodothyronine (Experimental)
  Interventions: Drug: Triiodothyronine; Drug: Sertraline
- sertraline + placebo (Placebo Comparator)
  Interventions: Other: Placebo; Drug: Sertraline

INTERVENTIONS:
Drug: Triiodothyronine
  Other Names: Cytomel
  Arms: sertraline + triiodothyronine
Other: Placebo
  Arms: sertraline + placebo
Drug: Sertraline
  Other Names: Zoloft

SUMMARY:
This study will evaluate the effectiveness of treatment with supplemental triiodothyronine (T3, Cytomel) and sertraline (Zoloft), a selective serotonin reuptake inhibitor (SSRI), in improving symptoms of major depressive disorder (MDD).

DETAILED DESCRIPTION:
The primary hypothesis is that triiodothyronine (Cytomel) supplementation of the antidepressant sertraline (Zoloft) will result in a greater improvement in HAM-D scores compared to placebo in the treatment of Major Depressive Disorder (MDD).

The goals of this proposal are to examine the relationship between Major Depressive Disorder (MDD) and abnormalities of the hypothalamic pituitary thyroid (HPT) axis. This protocol will systematically examine the value of supplemental triiodothyronine (T3, Cytomel) with sertraline (Zoloft), a selective serotonin reuptake inhibitor (SSRI) in the treatment of MDD. The focus will be on two overlapping populations: 1) those with evidence of HPT abnormalities, and 2) those who did not respond to a previous adequate SSRI trial

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 60. (The upper age is limited to 60 because thyroid changes, including blunting of the TSH response to TRH occurs with age and can potentially confound the relationship between the HPT axis and MDD.)
* Primary diagnosis of unipolar Major Depressive Disorder
* HAM-D (21 item) score >18

Exclusion Criteria:

* Alcohol abuse or alcohol dependence within the past year.
* Psychoactive substance abuse or dependence within the past year.
* Clinical evidence of severe Personality Disorder that would make study participation and completion unlikely.
* ECT within the past 6 months.
* Grade I hypothyroidism defined as low thyroid hormone levels with an associated elevated TSH; hyperthyroidism defined as elevated thyroid hormone concentrations with a low TSH.
* Serious and unstable medical illnesses.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 1996-09; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
MADRS score

SECONDARY OUTCOMES:
CGI

CONTACTS AND LOCATIONS:
Overall Officials: Boadie W Dunlop, MD, MS, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Result] Garlow SJ, Dunlop BW, Ninan PT, Nemeroff CB. The combination of triiodothyronine (T3) and sertraline is not superior to sertraline monotherapy in the treatment of major depressive disorder. J Psychiatr Res. 2012 Nov;46(11):1406-13. doi: 10.1016/j.jpsychires.2012.08.009. Epub 2012 Sep 7. PMID 22964160